CLINICAL TRIAL: NCT06689995
Title: An Investigation of the Safety and Effectiveness of an Oral Supplementation of Bio-Immune® for Managing Upper Respiratory Tract Infection and Its Symptoms: A Prospective, Interventional, Randomised, Double-Blind, Placebo-Controlled, Proof-of-Science Study.
Brief Title: A Clinical Study to Determine the Safety and Efficacy of an Oral Supplementation of Bio-Immune®for Managing Upper Respiratory Tract Infection and Its Symptoms.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Ambe Phytoextracts Pvt. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NB240047-AP
Record Dates: First submitted 2024-10-23; First posted 2024-11-15 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Upper Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-immune Capsule (Experimental): Dosage Form: Capsule Route of administration: Oral Frequency: 1 capsule, twice a day after meal for 5 days Dose: 100 mg
  Interventions: Other: Bio-immune Capsule
- Placebo Capsule (Placebo Comparator): Dosage Form: Capsule Route of administration: Oral Frequency: 1 capsule, twice a day after meal for 5 days Dose: 100 mg
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Bio-immune Capsule — Dosage Form: Capsule Route of administration: Oral Frequency: 1 capsule, twice a day after meal for 5 days Dose: 100 mg
  Arms: Bio-immune Capsule
Other: Placebo — Dosage Form: Capsule Route of administration: Oral Frequency: 1 capsule, twice a day after meal for 5 days
  Arms: Placebo Capsule

SUMMARY:
This is a prospective, interventional, randomised, double-blind, placebo-controlled, proof-of-science, in-use safety and efficacy study of an oral supplementation of Bio-Immune® for managing upper respiratory tract infection and its symptoms.

DETAILED DESCRIPTION:
A total of 54 human adults (27/arm) aged 30-80 years with uncomplicated Upper Respiratory Tract Infection will be enrolled to ensure the completion of 50 subjects (25/arm).

Potential subjects will undergo screening based on predefined inclusion and exclusion criteria only after obtaining written informed consent. The subject recruitment department will contact the potential subjects via telephone before the enrolment visit to confirm their participation.

Subjects shall be instructed to visit the facility for the following scheduled visits:

* Visit 1 [within 2 days]: Screening, evaluations for inclusion.
* Visit 2 [Day 1]: Enrolment, baseline and post-baseline evaluations, treatment commencement.
* Visit 3 [Day 2]: Test treatment usage phase, follow-up evaluations.
* Visit 4 [Day 3]: Test treatment usage phase, follow-up evaluations.
* Visit 5 [Day 5 (+1 day)]: End-of-study visit, follow-up Evaluations.

ELIGIBILITY:
Inclusion Criteria:

* 1. The age of subject is ≥30 years and <80 years. 2. The subject is a healthy male or a healthy adult non-pregnant and non-lactating female.

  3. The subject is suffering from uncomplicated URTI characterized by symptoms such as cough, nasal discharge, sore throat, or has had the first fever spike within 48 hours of enrolment.

  4. The subject must be willing to comply with all study procedures and restrictions, including taking the test treatment as directed, completing the WURSS-21 questionnaire, and undergoing laboratory assessments.

  5. The subject must provide written informed consent prior to participation in the study.

  6. The subject is in a stable medical condition, not requiring immediate intervention or hospitalization.

  7. If the subject is female, she is willing to use a highly effective method of contraception throughout the clinical investigation.
  1. Females of childbearing potential must practice and maintain an established method of birth control (e.g., IUD, hormonal implant device/injection, birth control pills, diaphragm, condoms with spermicide, partner vasectomy, or abstinence).
  2. Non-childbearing potential females who are surgically sterile, post-menopausal for at least 1 year, or have had a tubal ligation, must have been using hormonal contraception for at least 6 months and agree to continue using the same contraception for the study duration.

     Exclusion Criteria:
* 1. The subject is currently diagnosed with active respiratory infections or diseases other than uncomplicated URTI that might require immediate medical attention or intervention will be excluded.

  2. The chest X-ray of the subject, performed within the past 28 days, reveals significant respiratory disorders or other serious conditions that might interfere with the study or necessitate medical intervention.

  3. Laboratory tests (blood and urinalysis) performed at the screening visit reveal significant infective or other serious conditions that could interfere with the study or necessitate medical intervention.

  4. The subject has known immunocompromising conditions such as HIV/AIDS, or those undergoing immunosuppressive therapy.

  5. The subject has other significant respiratory diseases (e.g., COPD, asthma, interstitial lung disease, active tuberculosis).

  6. The subject has uncontrolled or severe cardiovascular, renal, or hepatic conditions.

  7. The subject has participated in any other clinical trial within 30 days prior to the screening visit.

  8. The subject is pregnant/lactating, or is planning on become pregnant during the course of the study.

  9. The subject has known hypersensitivity or allergies to any component of the test treatment or similar botanical extracts are excluded.

  10. The subject is on regular medications known to interfere with the study outcomes (e.g., systemic corticosteroids, antiviral drugs) within 4 weeks before screening are excluded.

  11. The subject has any condition that, in the investigator's judgment, would compromise the subject's safety or study integrity.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
To assess the effect of the test treatment on symptom severity and functional impairment scores as measured by the Wisconsin Upper Respiratory Symptom Survey-21 (WURSS-21) questionnaire, compared to placebo | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  Each symptom is rated on a 7-point scale, where "0" denotes "no symptom" and "7" denotes "severe symptoms."
To assess the effect of the test treatment on the overall symptom burden of the common cold, as determined by the Area Under the Curve (AUC) for the WURSS-21 symptom, functional impairment, and global scores, compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  Each symptom is rated on a 7-point scale, where "0" denotes "no symptom" and "7"

SECONDARY OUTCOMES:
To assess the effect of the test treatment on symptoms (such as cough), using a Visual Analogue Scale (VAS), compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  VAS which indicates 0: No Symptoms and 100: Worst Imaginable Symptoms
To assess the effect of the test treatment on symptoms (such as expectoration), using a Visual Analogue Scale (VAS), compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  VAS which indicates 0: No Symptoms and 100: Worst Imaginable Symptoms
To assess the effect of the test treatment on symptoms (such as nasal discharge), using a Visual Analogue Scale (VAS), compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  VAS which indicates 0: No Symptoms and 100: Worst Imaginable Symptoms
To assess the effect of the test treatment on symptoms (such as headache), using a Visual Analogue Scale (VAS), compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  VAS which indicates 0: No Symptoms and 100: Worst Imaginable Symptoms
To assess the effect of the test treatment on symptoms (such as fever), using a Visual Analogue Scale (VAS), compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  VAS which indicates 0: No Symptoms and 100: Worst Imaginable Symptoms
To assess the effect of the test treatment on symptoms (such as sore throat), using a Visual Analogue Scale (VAS), compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  VAS which indicates 0: No Symptoms and 100: Worst Imaginable Symptoms
To assess the effect of the test treatment on symptoms (such as earache), using a Visual Analogue Scale (VAS), compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  VAS which indicates 0: No Symptoms and 100: Worst Imaginable Symptoms
To assess the effect of the test treatment on symptoms (such as malaise/fatigue), using a Visual Analogue Scale (VAS), compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  VAS which indicates 0: No Symptoms and 100: Worst Imaginable Symptoms
To assess the effect of the test treatment on symptoms (such as cough), using the Numeric Rating Scale (NRS) by clinical evaluation for each symptom, compared to placebo | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  NRS Scale Where is 0: No symptom and 10: Worst Imaginable Symptom
To assess the effect of the test treatment on symptoms (such as expectoration), using the Numeric Rating Scale (NRS) by clinical evaluation for each symptom, compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  NRS Scale Where is 0: No symptom and 10: Worst Imaginable Symptom
To assess the effect of the test treatment on symptoms (such as nasal discharge), using the Numeric Rating Scale (NRS) by clinical evaluation for each symptom, compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  NRS Scale Where is 0: No symptom and 10: Worst Imaginable Symptom
To assess the effect of the test treatment on symptoms (such as headache), using the Numeric Rating Scale (NRS) by clinical evaluation for each symptom, compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  NRS Scale Where is 0: No symptom and 10: Worst Imaginable Symptom
To assess the effect of the test treatment on symptoms (such as fever), using the Numeric Rating Scale (NRS) by clinical evaluation for each symptom, compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  NRS Scale Where is 0: No symptom and 10: Worst Imaginable Symptom
To assess the effect of the test treatment on symptoms (such as sore throat), using the Numeric Rating Scale (NRS) by clinical evaluation for each symptom, compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  NRS Scale Where is 0: No symptom and 10: Worst Imaginable Symptom
To assess the effect of the test treatment on symptoms (such as earache), using the Numeric Rating Scale (NRS) by clinical evaluation for each symptom, compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  NRS Scale Where is 0: No symptom and 10: Worst Imaginable Symptom
To assess the effect of the test treatment on symptoms (such as malaise/fatigue), using the Numeric Rating Scale (NRS) by clinical evaluation for each symptom, compared to placebo. | on Day 1 (before administration) for baseline and 6 hours post-dosage, and later on Day 2, Day 3, and Day 5
  NRS Scale Where is 0: No symptom and 10: Worst Imaginable Symptom
To assess the effect of the test treatment on daily nasal discharge in terms of nasal mucus weight measured using pre-weighed paper tissues, compared to placebo. | on Day 1 (before administration) for baseline, and later on Day 2, and Day 3
  nasal mucus weighing kit - pre-weighed tissues and plastic bags with zip-lock seals
To assess the safety of the test treatment | To assess the safety of the test treatment by monitoring the occurrence of any adverse events throughout the study period. During the duration of the study of 0 to 5 Days.
  To assess the safety of the test treatment by monitoring the occurrence of any adverse events throughout the study period.
To assess the safety of the test treatment by evaluating Serum Creatinine. | on Day 1 (before administration) for baseline, and post-dosage on Day 5
  To assess the safety of the test treatment based on changes in blood parameters, including Serum Creatinine
To assess the safety of the test treatment by evaluating SGPT | on Day 1 (before administration) for baseline, and post-dosage on Day 5
  To assess the safety of the test treatment based on changes in blood parameter, including SGPT
To assess the safety of the test treatment by evaluating SGOT | on Day 1 (before administration) for baseline, and post-dosage on Day 5
  To assess the safety of the test treatment based on changes in blood parameter, including SGOT
To assess the safety of the test treatment by evaluating lipid profile | on Day 1 (before administration) for baseline, and post-dosage on Day 5
  To assess the safety of the test treatment based on changes in blood parameter, including Lipid Profile
To assess the safety of the test treatment by evaluating RBS | on Day 1 (before administration) for baseline, and post-dosage on Day 5
  To assess the safety of the test treatment based on changes in blood parameter, including RBS
To assess the safety of the test treatment by evaluating uric acid | on Day 1 (before administration) for baseline, and post-dosage on Day 5
  To assess the safety of the test treatment based on changes in blood parameter, including Uric acid
To assess the safety of the test treatment by evaluating Urinalysis | on Day 1 (before administration) for baseline, and post-dosage on Day 5
  To assess the safety of the test treatment in terms of change in urine analysis via Lab test
To assess the effectiveness of the test treatment in altering C-reactive protein levels in blood. | on Day 1 (before administration) for baseline, and post-dosage on Day 5
  Effectiveness of the test treatment evaluated in altering C-reactive protein levels in blood.
To assess the effectiveness of the test treatment by evaluating nasal wash sample. | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To assess the effectiveness of the test treatment altering biomarkers including IL-8 in nasal wash sample
To assess the effectiveness of the test treatment by evaluating IgA. | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To assess the effectiveness of the test treatment altering biomarkers including IgA in nasal wash sample, compared to placebo
To evaluate the safety of test treatment by evaluating Haemoglobin | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in Haemoglobin lab test
To evaluate the safety of test treatment by evaluating Haematocrit | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in Haematocrit using lab test
To evaluate the safety of test treatment by evaluating RBC Count | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in RBC Count using lab test
To evaluate the safety of test treatment by evaluating PCV Count | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in PCV Count using lab test
To evaluate the safety of test treatment by evaluating RBC Morphology | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in RBC Morphology using lab test
To evaluate the safety of test treatment by evaluating mean corpuscular volume (μm3) | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in mean corpuscular volume using lab test
To evaluate the safety of test treatment by evaluating Mean corpuscular haemoglobin (picograms (pg) per cell) | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in Mean corpuscular haemoglobin (picograms (pg) per cell)
To evaluate the safety of test treatment by evaluating Mean corpuscular hemoglobin concentration (g/dl) | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in Mean corpuscular hemoglobin concentration
To evaluate the safety of test treatment by evaluating red cell distribution width (%) | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in red cell distribution width
To evaluate the safety of test treatment by evaluating Total White Blood Cell Count (microliter ) | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in Total WBC Count using lab test
To evaluate the safety of test treatment by evaluating Differential WBC Count | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in Differential WBC Count usinglab test
To evaluate the safety of test treatment by evaluating Platelet Count | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in Platelet Count using lab test
To evaluate the safety of test treatment by evaluating mean platelet volume | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in mean platelet volume using lab test
To evaluate the safety of test treatment by evaluating Procalcitonin | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in Procalcitonin using blood test
To evaluate the safety of test treatment by evaluating Platelet distribution width | on Day 1 (before administration) for baseline, and post-dosage on Day 3
  To evaluate the safety of test treatment by evaluating change in Platelet distribution width using lab test

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Pvt.Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No